CLINICAL TRIAL: NCT04255849
Title: Nine-valent HPV Vaccine to Prevent Persistent Oral HPV Infection in Men Living With HIV
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other); University of Sao Paulo (Other); University of Puerto Rico (Other); National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry); University of California, San Diego (Other); Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19-11021038; U54CA242639 (NIH)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: HPV Positive Oropharyngeal Squamous Cell Carcinoma; HIV-1-infection; HPV Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 9-valent HPV vaccine (Experimental): Participants receive 9-valent HPV vaccine 0.5mL at entry, Month 2 and Month 6
  Interventions: Biological: 9 valent human papillomavirus vaccine (Types 6, 11, 16, 18, 31, 33, 45, 52, 58)
- Saline Placebo (Placebo Comparator): Participants receive 0.9% NaCl 0.5 mL at entry, Month 2 and Month 6
  Interventions: Other: Saline Placebo

INTERVENTIONS:
Biological: 9 valent human papillomavirus vaccine (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) — Gardasil-9 HPV vaccine
  Arms: 9-valent HPV vaccine
Other: Saline Placebo — Saline Placebo
  Arms: Saline Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled Phase III interventional trial of the nine-valent HPV vaccine (9vHPV) to prevent persistent oral HPV infection in adult men living with HIV.

DETAILED DESCRIPTION:
Men ages 20-50 years living with HIV will be enrolled at affiliated clinical sites of the University of Puerto Rico, the National Institute of Public Health, Mexico, and University of São Paulo, Brazil. Participants will have a baseline blood draw for serum HPV antibodies and stored plasma, an oral rinse for HPV testing, HPV methylation, and EBV co-infection, stored anal and genital samples for HPV testing, as well as a baseline questionnaire about risk factors for oral HPV infection and oropharyngeal cancer.

Seven hundred participants will be randomized in a 1:1 allocation to receive 9vHPV or placebo at Day 1, Month 2, and Month 6. Randomization will be stratified based on clinical site and age (20-30, 31-40, 41- 50 years). The age range of enrolled participants will be monitored to ensure enrollment of an approximately even distribution of participants across the age range. Enrollment will take place during the first 28 months of this study.

Follow-up testing for oral HPV will be conducted at Months 2, 6, 7, 12 and every 6 months thereafter up to 54 months post-vaccination. The rationale for oral testing at Months 2 and 6 is to identify participants who are oral HPV positive prior to receiving the full 3 doses of vaccine. In addition, an optional collection of anal canal and genital specimens (penile head, shaft, scrotum) will occur at Day 1, Months 7, 12 and every 6 months thereafter up to 54 months post-vaccination in those that specifically provided consent. These specimens will be stored for future medical research and will not be analyzed as part of this study. Serum will be stored for HPV antibody testing at month 7, 12 and every 12 months thereafter. Additionally, 20ml of whole blood will be collected beginning at Month 12 and every 12 months thereafter for DNA methylation of biological aging and circulating tumor HPV DNA (ctHPVDNA) analysis. Participants will undergo a follow-up questionnaire on risk factors for oral HPV and oropharyngeal cancer. Participants will be assessed for adverse events at each follow-up visit. This is a 5-year study. Participants who received placebo will be offered 9vHPV vaccine when the study is unblinded.

The trial analyses will be case driven with case counting commencing at Month 7, one month post-dose 3. The primary analysis will take place when at least 14 cases of the primary endpoint (incident persistent oral HPV infection with HPV types 6, 11, 16, 18, 31, 33, 45, 52, or 58) have been observed.

Early data on the baseline oral HPV prevalence among ULACNet-201 participants suggests an approximately 50% lower prevalence of oral HPV than anticipated. This suggests that oral HPV incidence will likely be significantly lower than anticipated. The reasons for this are not yet clear. To help speed the time until the required number of primary endpoint events is accrued, the number of events needed for the primary endpoint have been changed from 31 to 14. The sample size will also be increased by 40% (from 500 to 700 participants), of which a majority will be enrolled from sites in Mexico. Adding 200 participants will increase the number of follow-up visits where additional eligible primary endpoint events can occur. This allows for additional sample size should loss to follow-up increase. In addition, follow-up time will be extended from 42 months post-vaccination to 54 months post-vaccination to allow for accrual of at least 14 events.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Receipt of antiretroviral therapy for at least 6 months
* Sexually active in the past 6 months; sexual activity is defined as insertive penile-vaginal sex, receptive or insertive penile-anal sex, oral-anal sex, or oral-genital sex Willingness to comply with three-dose vaccine schedule and subsequent six-month visits for up to four years after randomization.

Exclusion Criteria:

* Have a history of oropharyngeal cancer (OPC) or other HPV-related cancer or have suspected OPC or other HPV-related cancer;
* Have received any doses of a licensed or experimental HPV vaccine or have participated in an HPV vaccine study,
* Have a history of anaphylaxis to vaccines or are allergic to any vaccine component (e.g.aluminum, yeast, benzonase);
* Have received any blood products within six months of enrollment, or are currently taking immune-suppressants.
* Currently have warts/lesions in the oral cavity.
* Plan to relocate during the study period.
* Have AIDS-defining condition within 6 months prior to study entry.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with new persistent oral HPV infections with one or more of the following types: 6, 11, 16, 18, 31, 33, 45, 52, or 58 | From Month 7 up to Month 60
  The primary endpoint is incident persistent oral HPV infection with HPV types 6, 11, 16, 18, 31, 33, 45, 52, or 58 occurring among participants who remain oral HPV negative to the relevant HPV type through the vaccination period (Day 1-Month 6). Newly acquired oral HPV infections that persist for two or more consecutive oral HPV assessments at least 16 weeks apart with the same 9vHPV detected are defined as "persistent". Case counting will commence with the Month 7 clinical visit and may occur at any timepoint through the final visit.

SECONDARY OUTCOMES:
Immunogenicity of 9-valent HPV vaccine as measured by proportion of participants experiencing seroconversion for vaccine type. | Month 7
  To evaluate our secondary immunogenicity endpoint, we will assess the proportion of men who seroconvert to the HPV vaccine types 6, 11, 16, 18, 31, 33, 45, 52, or 58 (both in grouped and type-specific analyses) in serum one month post-dose three (Month 7) using the Wilson's method. Men who enter the study seronegative for a particular HPV vaccine type will be monitored for seroconversion following three doses of 9vHPV.
Safety and tolerability of 9-valent HPV vaccine as measured by proportion of participants with >= grade 3 adverse events related to study vaccination or Grade 1 or 2 events leading to premature discontinuation of vaccination, or serious adverse events. | Baseline through Month 7
  To evaluate the secondary safety and tolerability endpoint, we will report the proportion of participants experiencing a grade 3 or 4 adverse event at least possibly related to study vaccine, grade 1 or 2 adverse events leading to premature discontinuation of vaccine or placebo, and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Ellsworth, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- Universidade de São Paulo, São Paulo, São Paulo, Brazil
- Instituto Nacional de Salud Pública, Mexico, Cuernavaca, Morelos, Mexico
- University of Puerto Rico AIDS Clinical Trials Unit, San Juan, Purto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months following publication and available through period of funding of ULACNet (U54 CA242639).
Access Criteria: Researchers who provide a methodologically sound proposal for use of the data that is approved by the study investigators and the sponsor.
  The research must be broadly consistent with that of ULACNet.
  Researchers may submit a request to the study principal investigator (Grant Ellsworth gre9006@med.cornell.edu) to request details of request format.

REFERENCES:
- [Derived] Giuliano AR, Beltrame A, Villa LL, Lazcano-Ponce E, Santana-Bagur J, Allen-Leigh B, Portillo-Romero AJ, Sahasrabuddhe VV, House MG, Brofsky E, Galan de Paula L, Carvalho da Silva R, Schell MJ, Rathwell J, Isaacs-Soriano K, Fan W, Mello C, Ellsworth GB, Wilkin T. Design of a multicenter, randomized, double-blinded, placebo-controlled phase III trial evaluating the 9-valent human papillomavirus (HPV) vaccine to prevent persistent oral HPV infection in men living with human immunodeficiency virus: ULACNet trial 201. Vaccine. 2025 Aug 13;61:127447. doi: 10.1016/j.vaccine.2025.127447. Epub 2025 Jul 2. PMID 40609265